CLINICAL TRIAL: NCT03487380
Title: Taxonomic and Functional Composition of the Intestinal Microbiome: a Predictor of Rapid Cognitive Decline in Patients With Alzheimer's Disease
Acronym: MiDCR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Despite an extension of the planned duration of inclusion and an enrolled patient number inferior than planned, coordinating investigator considered that it was more reasonable to stop inclusions in order to analyze the data already available
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC17_0162; 2017-A02246-47 (Other: ANSM)
Record Dates: First submitted 2018-03-27; First posted 2018-04-04 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Alzheimer Disease; Intestinal Microbiota
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The study will compare three groups of 100 patients, corresponding to 200 patients with Alzheimer disease (whom 100 patients in the rapid cognitive decline group and 100 patients without rapid cognitive decline) and 100 patients in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alzheimer with rapid DCR (Experimental)
  Interventions: Procedure: Fecal sample collection
- Alzheimer without rapid DCR (Experimental)
  Interventions: Procedure: Fecal sample collection
- Control (Sham Comparator)
  Interventions: Procedure: Fecal sample collection

INTERVENTIONS:
Procedure: Fecal sample collection — Fecal sample collection

SUMMARY:
The objective of the study is to highlight a modification of the composition of the intestinal microbiota associated with the diagnosis of Alzheimer's disease and its most unfavorable form, Rapid Cognitive Decline (DCR). This identification could lead to diagnostic strategies based on the analysis of the intestinal microbiome, and preventive and curative treatments, based on the modulation of intestinal microbiota

ELIGIBILITY:
Inclusion Criteria:

For Alzheimer groups without DCR and Alzheimer with DCR:

* patients between 70 and 90 years old
* with mild to moderate Alzheimer's disease (MMSE> 15/30),
* followed in the CMRR of the University Hospital of Nantes or Angers
* having given their informed consent

For the control group (non-Alzheimer's)

* more patients between 70 and 90 years
* consultant for a subjective memory complaint isolated at the CMRR of Nantes or Angers University Hospital,
* having given their informed consent

Exclusion Criteria:

* Major patients under tutorship, curatorship or safeguard of justice
* Cognitive disorders possibly related to a metabolic or psychiatric cause
* History of prescription of antibiotic treatment in the last month
* History of acute gastrointestinal illness in the last month
* History of hospitalization for an acute medical pathology or for a surgical procedure in the last month

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
analysis of the taxonomic and functional composition of the microbiome | 1 year
  ("shotgun sequencing"), in patients with DCR (loss of at least 3 points in the MMSE at 1 year.

SECONDARY OUTCOMES:
to determine if there is a specific modification of the composition of the intestinal microbiota of patients with Alzheimer's disease, compared to control group. | Day 0
create a prognostic score of DCR based on clinical data, including the responses to the MMSE, BREF and MNA questionnaires, and taking into account the microbiota analysis | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Angers, Angers
  - CHU de Nantes, Nantes